CLINICAL TRIAL: NCT04193943
Title: Validation Study of Simplified Electrophysiological Examination in the Diagnosis of Critical Illness Myopathy or Neuropathy
Brief Title: Validation of Simplified Electrophysiological Examination in the Diagnosis of Critical Illness Myopathy or Neuropathy
Acronym: CRIMINE-3
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Elisa Seghelini,MD, Principal Investigator, Università degli Studi di Brescia
Other Study IDs: PN 1700/2014
Record Dates: First submitted 2019-11-25; First posted 2019-12-11 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Critical Illness Polyneuropathy; Critical Illness Myopathy
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the accuracy, in the diagnosis of critical illness myopathy and / or neuropathy, of the simplified peroneal nerve test performed by a neurophysiopathology technician or by a neurophysiopathology doctor (as the gold standard) compared to the exam performed by an intensivist.

ELIGIBILITY:
Inclusion Criteria:

- adult patients admitted to Intensive care unit

Exclusion Criteria:

* patients in terminal conditions
* patients with peroneal nerve exam not feasible ( for example with presence of prostheses, wounds, plaster casts, edema of the limbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically Ill Patients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-06-18 (Actual); Primary Completion 2014-11-26 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of peroneal nerve test performed by a neurophysiopathologist compared to peroneal nerve test performed by an intensivist when peroneal nerve test is dichotomised in normal or abnormal | up to the comlpete execution of the two peroneal nerve exams,at most an hour
  DTComPair-package in R
specificity of peroneal nerve test performed by a neurophysiopathologist compared to peroneal nerve test performed by an intensivist when peroneal nerve test is dichotomised in normal or abnormal | up to the comlpete execution of the two peroneal nerve exams, at most an hour
  DTComPair-package in R

SECONDARY OUTCOMES:
evaluation of concordance between peroneal nerve test performed by an intensivist compared to peroneal nerve test performed by a neurophysiopathologist considering the test as a continuous variable | up to the comlpete execution of the two peroneal nerve exams, at most an hour
  It will be performed either using Bland-Altman plot and mix model effect
correlation between hospital mortality and abnormal peroneal nerve test | up to hospital discharge, an average of 6 months
  Anova
correlation between hospital discharge destination and abnormal peroneal nerve test | up to hospital discharge, an average of 6 months
  Anova

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Seghelini, Principal Investigator — II Servizio di Anestesia e Rianimazone, Spedali Civili
Locations (1):
- Spedali Civili, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No